CLINICAL TRIAL: NCT02334098
Title: Omega-3 Supplementation and Behavior Problems in Children and Adolescents
Brief Title: Omega-3 Supplementation and Behavior Problems
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Annis Fung (Other)
Collaborators: University of Pennsylvania (Other); The University of Hong Kong (Other); Brooklyn College of the City University of New York (Other)
Responsible Party: Sponsor-Investigator, Dr. Annis Fung, Associate Professor, City University of Hong Kong
Organization: City University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GRF-11402514
Record Dates: First submitted 2014-12-29; First posted 2015-01-08 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Aggression; Antisocial Behavior; Antisocial Personality
Keywords: Aggression; Omega-3 supplementation; Neurocognition; Attention; Antisocial
MeSH Terms: conditions — Aggression; Antisocial Personality Disorder

STUDY DESIGN:
Intervention Model Description: 3 parallel groups: (1) omega-3 + fruit juice (2) fruit juice only (3) controls (no drink).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: all participants and research assistants are blind to condition for the two fruit juice groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega-3 supplemented drink (Experimental): A 200 ml. drink product with 1.1 grams of omega-3 from Smartfish (Smartfish: Forsiden in Norway).
  Interventions: Dietary Supplement: Omega-3 supplemented drink
- Placebo Drink (Placebo Comparator): exactly the same fruit drink contained in the same packaging, but will contain no omega-3.
  Interventions: Dietary Supplement: Smartfish
- treatment-as-usual controls (No Intervention): No drinks are taken.

INTERVENTIONS:
Dietary Supplement: Omega-3 supplemented drink — The drink has apple/ pear/ pomegranate taste which is well accepted by children and adolescents, is rich in natural antioxidants to help prevent oxidation of omega-3. The drink can be taken at any time during the day.
  1/3 of the participants will be assigned to the omega-3 group after randomization. They are going to take the treatment for 6 months. They will be assessed at baseline, end of treatment and 6 months post-treatment.
  Arms: Omega-3 supplemented drink
Dietary Supplement: Smartfish — Treatment duration is 6 months. They will be assessed at baseline (0 months), end of treatment (6 months) and 6 months post-treatment (12 months).
  Arms: Placebo Drink

SUMMARY:
The objectives of this project are as follows:

1. To assess whether omega-3 dietary supplementation for six months can reduce externalizing behavior problems (antisocial and aggressive behavior) in schoolchildren aged 8 to 18, both at the end of treatment and six months post-treatment
2. To assess whether omega-3 supplementation is more effective in children with more psychopathic-like traits.

DETAILED DESCRIPTION:
Externalizing behavior problems (aggressive and antisocial behaviors) are widely recognized as predisposing to significant mental health problems and violence among adolescents in secondary schools. These in turn result in enormous economic and social costs to schools as well as to society. These costs include mental illness, crime, and violence. Similarly, violence is widely recognized as a major public health problem which has also largely defied successful intervention and prevention. Because an increasing body of research is documenting health and neurobiological risk factors for aggression and violence, part of this prevention failure may be due to intervention efforts ignoring biological contributory factors which include impaired neurocognitive and psychophysiological functioning. One benign biological intervention that may help attenuate behavior problems in children consists of omega-3 supplementation of the diet, a long-chain fatty acid critical for brain structure and function.

The overarching aim of this study is to assess whether omega-3 supplementation can reduce the base level of externalizing behavior problems in children and adolescents. A secondary but important aim is to assess whether any behavioral improvement may be greater in more psychopathic children. The specific aims are as follows:

1. To assess the effectiveness of omega-3 dietary supplementation in reducing externalizing behaviors in adolescents.
2. To assess whether omega-3 supplementation leads to greater improvement in children with psychopathic-like traits.

Hypotheses will be tested in a placebo-controlled, double-blind, randomized trial involving 8 to18 year-old adolescents drawn from primary and secondary schools in Hong Kong. Omega-3 supplementation will be in the form of a Norwegian fruit juice drink. 300 adolescents will be randomly assigned into: (1) omega-3 supplemented drink, (2) placebo drink, (3) treatment-as-usual controls. Behavioral measures will be assessed at baseline (0 months), end of treatment (6 months), and 6 months post-treatment (12 months).

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents between the age 8 and 18
* participants who does not fit in any of the following exclusion criteria

Exclusion Criteria:

* unwilling to participate in a randomized, double-blind, placebo controlled trial,
* unable to give written, informed parental consent and assent from children,
* on medication that may modify lipid metabolism in the past 3 months
* significant use of omega-3 supplements in the past 6 months
* seafood allergies
* mental retardation
* epilepsy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 324 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Externalizing and internalizing behavior problems | up to 12 months after initiation of trial: assessement at 0 months, 6 months (end of treatment) and 12 months (6 months post-tretament)
  The following instruments will be administered to both caregivers and the children to assess child behavior behavior problems (externalizing and internalizing)
  Adolescent self-reported measures include Reactive-Proactive Aggression Questionnaire (RPQ), Antisocial Personality Screening Device (APSD), Conduct and Oppositional Defiant Disorder Questionnaire (COD) and Child Behavior Checklist (CBCL - Attention and Anxiety/Depressed subscales only).

SECONDARY OUTCOMES:
Neurocognitive functioning | up to 12 months
  Neurocognitive functioning is assessed by the Tower of London. The Tower of London is an assessment tool to examine the functional anatomy of planning. It assesses high-order problem solving, specifically, executive planning abilities.
Psychophysiological functioning | up to 12 months
  Psychophysiological (attentional) functioning is assessed using EEG (P300 oddball task).
Emotional empathy | up to 12 months
  measured by a 10-items self-report instrument (CASES)
Grit | up to 12 months
  measured by an 8-item self-report instruments (GRIT)

CONTACTS AND LOCATIONS:
Overall Officials: Annis Fung, Ph.D., Principal Investigator — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, China